CLINICAL TRIAL: NCT00320398
Title: Clinical Evaluation of GSK576428 (Fondaparinux Sodium) in Prevention of Venous Thromboembolism After Elective Total Hip Replacement Surgery
Brief Title: Total Hip Replacement Study Of GSK576428 (Fondaparinux Sodium)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: AR3106333
Record Dates: First submitted 2006-05-01; First posted 2006-05-03 (Estimated); Results first posted 2017-12-21 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Thrombosis, Venous
Keywords: Fondaparinux; Hip Replacement Arthroplasty; VTE; THR; MOSLL; pentasaccharide; Xa factor
MeSH Terms: conditions — Venous Thrombosis | interventions — Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Fondaparinux

SUMMARY:
This study is requested by PMDA to confirm the optimal dose for THR (total hip replacement).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing either an elective primary THR (total hip replacement) surgery or a revision of a THR.

Exclusion Criteria:

* Active, clinically significant bleeding (excluding drainage).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2006-01-30 (Actual); Primary Completion 2006-07-18 (Actual); Study Completion 2006-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 115 participants who had undergone total Hip replacement surgery were randomized to the study. The study was conducted from 30 January 2006 to 18 July 2006 at eight centers in Japan. A total of 114 and 94 participants were included in Safety and Full analysis set population respectively.
Groups:
- Fondaparinux 1.5 mg: Eligible participants in this arm received fondaparinux at 1.5 milligram (mg) administered as a subcutaneous injection once daily for 10 to 14 days (between Day 2 and Day 11- 15), (where Day 1 was the day of surgery). The first injection of the study drug was given 24 + or - 2 hours after the surgical closure. From Day 3 onwards the injection of the study drug was given at about the same time every day as far as possible (but more than 12 hours after the first dose on Day 2).
- Fondaparinux 2.5 mg: Eligible participants in this arm received fondaparinux at 2.5 mg, administered as a subcutaneous injection once daily for 10 to 14 days (between Day 2 and Day 11- 15), (where Day 1 was the day of surgery). The first injection of the study drug was given 24 + or - 2 hours after the surgical closure. From Day 3 onwards the injection of the study drug was given at about the same time every day as far as possible (but more than 12 hours after the first dose on Day 2).
Period: Overall Study
Arm/Group | Fondaparinux 1.5 mg | Fondaparinux 2.5 mg
Started | 58 | 56
Completed | 56 | 52
Not Completed | 2 | 4
Not completed — Adverse Event | 1 | 4
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fondaparinux 1.5 mg: Eligible participants in this arm received fondaparinux at 1.5 mg, administered as a subcutaneous injection once daily for 10 to 14 days (between Day 2 and Day 11- 15), (where Day 1 was the day of surgery). The first injection of the study drug was given 24 + or - 2 hours after the surgical closure. From Day 3 onwards the injection of the study drug was given at about the same time every day as far as possible (but more than 12 hours after the first dose on Day 2).
- Total: Total of all reporting groups
Arm/Group | Fondaparinux 1.5 mg | Fondaparinux 2.5 mg | Total
Number analyzed (Participants) | 58 | 56 | 114
Age, Customized [Count of Participants; unit: Participants]
  >=20 years | 58 | 56 | 114
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 51 | 102
  Male | 7 | 5 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 58 | 56 | 114

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Venous Thromboembolism (VTE) During Efficacy Period
Description: The percentage of participants with VTE, who underwent elective total hip replacement surgery, detected by routine venography, during the treatment period were reported. The percentage VTE was calculated by the number of events divided by the number of participants evaluated multiplied by 100. The Venogram was obtained post 2 calendar days after the administration of last study drug (between Day 11 and 17). Day 1 was the day of surgery and the participant was given study drug 24±2 hours after surgical closure. It was adjudicated by the Central Independent Adjudication Committee of Efficacy (CIACE).
Time Frame: Up to Day 17
Population: The Full Analysis Set (FAS) population consisted of all participants who were randomized to either treatment with the exception of: those who did not receive study drug at all; and those with no valid post-randomization efficacy data (e.g., no evaluable venogram).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fondaparinux 1.5 mg | Fondaparinux 2.5 mg
Number analyzed (Participants) | 48 | 46
percentage of participants | 8.3 [2.3 to 20.0] | 2.2 [0.1 to 11.5]

2. Primary Outcome: Percentage of Participants With Major Bleeding
Description: Major bleeding defined as any clinically unusual bleeding meeting 1 of following criteria; a)Fatal bleeding; b) Including retroperitoneal and intracranial bleeding, or bleeding into critical organ (eye, adrenal gland, pericardium, spine); c) Reoperation due to bleeding or hematoma at operative site; d)Bleeding leading to hemoglobin (Hb) fall > = 2 gram per deciliter (g/dL)(1.6 millimole per litre [mmol/L]) within 48 hour of the bleed; e)Bleeding that required transfusion of red blood cells (RBCs) or whole blood (WB) derived from >= 900 milliliter (mL) of WB within 48 hours of the bleed (excluding autologous transfusion except for treatment of bleeding adverse event); f) Bleeding leading to bleeding index (BI) >=2. The percentage was calculated by the number of events divided by the number of participants evaluated multiplied by 100. This was adjudicated by the CIACE.
Time Frame: Up to Day 17
Population: The safety population consisted of all participants who received at least one dose of randomized study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fondaparinux 1.5 mg | Fondaparinux 2.5 mg
Number analyzed (Participants) | 58 | 56
percentage of participants | 0 [0.0 to 6.2] | 0 [0.0 to 6.4]

3. Secondary Outcome: Percentage of Participants With Minor Bleeding
Description: Minor bleeding was defined as the clinically overt bleeding not meeting the criteria for major bleeding like: (Fatal bleed; Including retroperitoneal and intracranial bleeding, or bleed in critical organ [eye, adrenal gland, pericardium, spine]; c) Reoperation due to bleeding or hematoma at operative site; d) Bleeding leading to hemoglobin (Hb) fall > = 2 g/dL(1.6 mmol/L) within 48 hour of the bleed; e)Bleeding that required transfusion of RBCs or WB derived from >= 900 mL of WB within 48 hours of the bleed (excluding autologous transfusion except for treatment of bleeding adverse event); f) Bleeding leading to bleeding index (BI) >=2), and which were considered more than expected in the clinical context. The percentage was calculated by the number of events divided by the number of participants evaluated multiplied by 100. This was adjudicated by the CIACE.
Time Frame: Up to Day 17
Population: Safety population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fondaparinux 1.5 mg | Fondaparinux 2.5 mg
Number analyzed (Participants) | 58 | 56
percentage of participants | 1.7 [0.0 to 9.2] | 3.6 [0.4 to 12.3]

4. Secondary Outcome: Percentage of Participants With All Deep Vein Thrombosis (DVT)
Description: The percentage of participants with All DVT were reported, where the analysis was done using a venogram. It was calculated by the number of events divided by the number of participants evaluated multiplied by 100. The Venogram was obtained post 2 calendar days after the administration of last study drug (between Day 11 and 17). Day 1 was the day of surgery and the participant was given study drug 24±2 hours after surgical closure. It was adjudicated by the CIACE.
Time Frame: Up to Day 17
Population: Efficacy Evaluable Patients (EEP) included subpopulation of safety participants judged to be evaluable for all DVT, proximal DVT or distal only DVT by site of occurrence (total/ side of operation/ opposite side of operation/ both sides). Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Fondaparinux 1.5 mg | Fondaparinux 2.5 mg
Number analyzed (Participants) | 48 | 46
percentage of participants | 8.3 | 2.2

5. Secondary Outcome: Percentage of Participants With Proximal DVT
Description: The percentage of participants with DVT (proximal) were reported, by using a venogram. It was calculated by the number of events divided by the number of participants evaluated multiplied by 100. The Venogram was obtained post 2 calendar days after the administration of last study drug (between Day 11 and 17). Day 1 was the day of surgery and the participant was given study drug 24±2 hours after surgical closure. It was adjudicated by the CIACE.
Time Frame: Up to Day 17
Population: EEP population. Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Fondaparinux 1.5 mg | Fondaparinux 2.5 mg
Number analyzed (Participants) | 53 | 52
percentage of participants | 0 | 0

6. Secondary Outcome: Percentage of Participants With Distal Only DVT
Description: The percentage of participants with distal only DVT were reported, by using a venogram. It was calculated by the number of events divided by the number of participants evaluated multiplied by 100. The Venogram was obtained post 2 calendar days after the administration of last study drug (between Day 11 and 17). Day 1 was the day of surgery and the participant was given study drug 24±2 hours after surgical closure. It was adjudicated by the CIACE.
Time Frame: Up to Day 17
Population: EEP population. Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: percentage participants
Groups:
- Fondaparinux 1.5 mg: Eligible participants in this arm received fondaparinux at 1.5 mg administered as a subcutaneous injection once daily for 10 to 14 days (between Day 2 and Day 11- 15), (where Day 1 was the day of surgery). The first injection of the study drug was given 24 + or - 2 hours after the surgical closure. From Day 3 onwards the injection of the study drug was given at about the same time every day as far as possible (but more than 12 hours after the first dose on Day 2).
Arm/Group | Fondaparinux 1.5 mg | Fondaparinux 2.5 mg
Number analyzed (Participants) | 48 | 46
percentage participants | 4 | 1

7. Secondary Outcome: Percentage of Participants With Symptomatic DVT During Main Efficacy Period
Description: The percentage of participants with different symptoms of DVT (proximal) like pain or tenderness, swelling, warmth, redness or discoloration, and distention of surface veins, post the total hip replacement surgery were reported, where analysis was done using a venogram. It was calculated by the number of events divided by the number of participants evaluated multiplied by 100. The Venogram was obtained post 2 calendar days after the administration of last study drug (between Day 11 and 17). Day 1 was the day of surgery and the participant was given study drug 24±2 hours after surgical closure. It was adjudicated by the CIACE.
Time Frame: Up to Day 17
Population: Safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Fondaparinux 1.5 mg | Fondaparinux 2.5 mg
Number analyzed (Participants) | 58 | 56
percentage of participants | 0 | 0

8. Secondary Outcome: Percentage of Participants With Pulmonary Embolism During Efficacy Period
Description: The percentage of participants with pulmonary embolism (pleuritic chest pain, dyspnea, cough, hemoptysis, syncope, light-headedness/dizziness, tachypnea, and tachycardia ) were reported, by using a venogram. It was calculated by the number of events divided by the number of participants evaluated multiplied by 100. The Venogram was obtained post 2 calendar days after the administration of last study drug (between Day 11 and 17). Day 1 was the day of surgery and the participant was given study drug 24±2 hours after surgical closure. It was adjudicated by the CIACE.
Time Frame: Up to Day 17
Population: Safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Fondaparinux 1.5 mg | Fondaparinux 2.5 mg
Number analyzed (Participants) | 58 | 56
percentage of participants | 0 | 0

9. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Deaths
Description: An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. For marketed medicinal products, this also includes failure to produce expected benefits (i.e. lack of efficacy), abuse or misuse. SAE was any experience that: resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was medically significant.
Time Frame: From first injection of study drug (Day 3) to up to 2 calendar days after last injection (Treatment period), up to Day 17.
Population: Safety population.
Measure: Number; unit: participants
Arm/Group | Fondaparinux 1.5 mg | Fondaparinux 2.5 mg
Number analyzed (Participants) | 58 | 56
participants
  Deaths | 0 | 0
  Any SAE | 0 | 0
  Any AE | 49 | 45

10. Secondary Outcome: Number of Transfused Participants
Description: The number of participants who received RBCs or WB after the total hip replacement surgery within 48 hours of bleed were reported.
Time Frame: Up to Day 17.
Population: Safety population.
Measure: Number; unit: participants
Arm/Group | Fondaparinux 1.5 mg | Fondaparinux 2.5 mg
Number analyzed (Participants) | 58 | 56
participants | 5 | 2

11. Secondary Outcome: Volume of Transfusion
Description: The total volume of transfusion (RBCs or WB) received by the participant was reported.
Time Frame: Up to Day 17
Population: Safety population.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Fondaparinux 1.5 mg | Fondaparinux 2.5 mg
Number analyzed (Participants) | 58 | 56
mL | 400.0 (0.0) | 600.0 (282.8)

ADVERSE EVENTS:
Time Frame: From first injection of study drug (Day 3) to up to 2 calendar days after last injection (Treatment period), up to Day 17.
Description: Safety population was used.
Arm/Group | Fondaparinux 1.5 mg | Fondaparinux 2.5 mg
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/56
Other Adverse Events (participants affected / at risk) | 49/58 | 45/56
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fondaparinux 1.5 mg (N=58) | Fondaparinux 2.5 mg (N=56)
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 14
Insomnia (Psychiatric disorders) | 9 | 13
Constipation (Gastrointestinal disorders) | 5 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 9
Platelet count increased (Investigations) | 7 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4
Gamma glutamyl transferase increased (Investigations) | 1 | 3
Headache (Nervous system disorders) | 5 | 2
Dizziness (Nervous system disorders) | 3 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 2 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Pyrexia (General disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.